CLINICAL TRIAL: NCT04100525
Title: Neuropsychological Feedback Style and Case Management to Improve Intervention Outcome for Employed Women With Multiple Sclerosis: a Randomized Clinical Trial
Brief Title: Intervention for Employed Women With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Holy Name Medical Center, Inc. (Other)
Collaborators: Women United in Philanthropy (WUIP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Employment Study
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: Employment; Vocational Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were informed that they would receive feedback but were not told whether it would be in person or by phone until after randomization. Participants were not informed that only one group received case management calls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Participant received neuropsychological testing, report detailing cognitive strengths and weaknesses, tailored recommendations to address areas of weakness (including psychological and/or physical symptoms impacting work productivity). Participant received a copy of this report in the mail and a call from the psychologist to go over test findings and recommendations.
  Interventions: Behavioral: Neuropsychological testing intervention plus follow up
- Experimental Treatment (Experimental): Participant received neuropsychological testing, report detailing cognitive strengths and weaknesses, tailored recommendations to address areas of weakness (including psychological and/or physical symptoms impacting work productivity). Participant then receives in-person feedback (and a copy of the report at this visit) and two calls from a care-coordinator research nurse at approximately 1 and 6 months post feedback, who asks participant whether they completed recommendations and assist participant in completing recommendations where possible (i.e., help find a provider, explanation of importance of completing recommendations, etc).
  Interventions: Behavioral: Neuropsychological testing intervention plus follow up

INTERVENTIONS:
Behavioral: Neuropsychological testing intervention plus follow up — Neuropsychological testing for women experiencing significant fatigue, mood, or cognitive symptoms. Feedback type and case management services varied depending on randomized group.

SUMMARY:
Unemployment is particularly common among women with multiple sclerosis (MS). This study uses a vocational rehabilitation program involving neuropsychological testing as an intervention. The use of in-person feedback and case management following neuropsychological testing is compared to phone feedback only. Adherence to treatment and employment outcomes will be evaluated over three years.

DETAILED DESCRIPTION:
Employed women at a tertiary-care MS center were screened for common issues impacting work productivity (fatigue, cognitive dysfunction, and depression). Women who met screening criteria were randomized to one of two treatment groups: either neuropsychological testing and phone feedback to review findings and tailored recommendations (standard-care treatment); or neuropsychological testing, in-person feedback, and two calls from a care-coordinator (experimental treatment). Adherence to recommendations and employment status at one year are evaluated. Follow-up periods also occur at year two and year three.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age between 18 and 64
* Employed at least 20 hours per week
* Confirmed diagnosis of MS

Exclusion Criteria:

* Experiencing an MS exacerbation
* Endorsing suicidal ideation or intent
* Pregnant
* Severe psychiatric disorder
* History of traumatic brain injury
* Dementia
* Major neurological illness other than MS

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study targeted females
Enrollment: 89 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Employment | Approximately 12 months
  Has there been a decrease in employment status (Yes/No)

SECONDARY OUTCOMES:
Adherence to Recommendations | Approximately 12 months
  Percentage of recommendations completed at one year

CONTACTS AND LOCATIONS:
Overall Officials: Frederick W Foley, Ph.D., Principal Investigator — Holy Name Medical Center, Ferkauf Graduate School of Psychology

IPD SHARING:
Plan to Share IPD: No